CLINICAL TRIAL: NCT01754324
Title: The Utility and Pharmacokinetics of Oral Methadone in the Treatment of Neonatal Abstinence Syndrome in Neonates
Brief Title: The Pharmacokinetics of Oral Methadone in the Treatment of Neonatal Abstinence Syndrome
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jason Wiles, MD, Neonatology Fellow, Children's Hospital Medical Center, Cincinnati
Other Study IDs: CCHMC-PK-1; 5T32HD069054 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-21 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Neonatal Abstinence Syndrome; Pharmacokinetics; Methadone; Neonate; Newborn
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Methadone: All infants requiring pharmacological treatment of their NAS symptoms are treated with a standardized protocol utilizing oral methadone. This treatment protocol has been the standard of care for infants with NAS at our institution for many years. Infants enrolled in this study will have blood samples drawn at predetermined times in order to obtain information regarding the pharmacokinetics of oral methadone in this population.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — The starting dose of the protocol is 0.05mg/kg by mouth given every 6 hours and gradually decreased in a stepwise, standardized fashion.
  Other Names: methadone hydrochloride

SUMMARY:
The chronic use of opiate medications during pregnancy is a major public health challenge. Prolonged exposure to opiates in utero may result in withdrawal symptoms in infants commonly referred to as neonatal abstinence syndrome (NAS). Signs of NAS may include irritability, high-pitched crying, muscle tightness, seizures, diarrhea, vomiting, poor feeding, and unstable body temperature. Many infants may be treated by supportive (non-pharmacological) therapy by minimizing stimulation, cuddling, responding promptly to hunger cues, and other comfort care. However, some infants continue to show severe symptoms of withdrawal despite these interventions. In these cases, infants may be treated with medications (pharmacological therapy). Although it has been several decades since the first descriptions of NAS, there still remains limited information with regards to the most effective treatment. We hypothesize that medical treatment protocols of NAS with methadone can be optimized by better understanding what the body does to the drug (the population-based pharmacokinetics of methadone).

ELIGIBILITY:
Inclusion Criteria:

1. Chronic in utero exposure to opiates
2. Term infant, greater than or equal to 37 weeks gestation
3. Failure of non-pharmacologic treatment of NAS
4. Infant meets criteria for pharmacologic treatment of NAS as determined by physical findings consistent with drug withdrawal and Finnegan scoring system
5. The attending neonatologist chooses to treat the qualifying infant with oral methadone.

Exclusion Criteria:

1. Prematurity
2. Congenital Abnormalities
3. Acutely ill neonates
4. Confounding medical illness necessitating therapy with opiates other than for NAS
5. Neonates whose only exposure to opiates were narcotics administered during labor
6. Infants who are wards of the state

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants diagnosed with Neonatal Abstinence Syndrome and are treated with oral methadone.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Methadone and EDDP (2-ethylidene-1,5-dimethyl-3,3-diphenylpyrrolidine) blood concentration | Participants will be followed for the duration of the hospital stay (an expected average of 4 weeks).
  Timed blood samples will be collected to estimate pharmacokinetic parameters of oral methadone and its major metabolite EDDP using population pharmacokinetic methods.

SECONDARY OUTCOMES:
Failed Protocol Wean | Participants will be followed for the duration of the hospital stay (an expected average of 4 weeks).
  Blood specimens for the analysis of methadone and EDDP concentrations will be obtained from infants who do not tolerate the standard methadone dosing taper to investigate its utility in identifying rapid metabolizers of methadone.
Number of participants requiring adjunctive pharmacological treatment | Participants will be followed for the duration of the hospital stay (an expected average of 4 weeks).
  This endpoint will look at the number of patients who require supplemental phenobarbital in the treatment of NAS symptoms.
Length of hospitalization | Participants will be followed for the duration of the hospital stay (an expected average of 4 weeks).
  This endpoint will describe the number of days infants were hospitalized for treatment of NAS.
Readmission to the hospital | Participants will be followed for the duration of the hospital stay (an expected average of 4 weeks) and will complete a follow-up survey up to 2 weeks after hospital discharge.
  This endpoint will describe the number of infants treated for NAS who later developed withdrawal symptoms after discharge that required readmission to the hospital.
Clinical resolution of NAS symptoms | Participants will be followed for the duration of the hospital stay (an expected average of 4 weeks) and will complete a follow-up survey up to 2 weeks after hospital discharge.
  The length of medical therapy with oral methadone (in days) required to result in the clinical resolution of NAS symptoms will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Wiles, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Henry Akinbi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Alexander Vinks, PharmD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - The University Hospital, Cincinnati, Ohio
  - Mercy Hospital Anderson, Cincinnati, Ohio

REFERENCES:
- [Derived] Wiles JR, Isemann B, Mizuno T, Tabangin ME, Ward LP, Akinbi H, Vinks AA. Pharmacokinetics of Oral Methadone in the Treatment of Neonatal Abstinence Syndrome: A Pilot Study. J Pediatr. 2015 Dec;167(6):1214-20.e3. doi: 10.1016/j.jpeds.2015.08.032. Epub 2015 Sep 11. PMID 26364984